CLINICAL TRIAL: NCT01899300
Title: A Multi-Center, Prospective, Evaluation of the Use of a Fully Covered Metal Stent (FCMS) for the Treatment of Refractory Benign Esophageal Strictures Caused by Caustic Ingestion
Brief Title: Esophageal Fully Covered Metal Stents in Caustic Strictures Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 90871111
Record Dates: First submitted 2013-06-28; First posted 2013-07-15 (Estimated); Results first posted 2021-02-12 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2021-01

CONDITIONS: Refractory Benign Esophageal Strictures Caused by Caustic Ingestion
Keywords: Refractory Benign Esophageal Strictures caused by Caustic Ingestion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Metal Stent (Experimental): The WallFlex™ Esophageal Fully Covered Metal Stent (FCMS)is being evaluated for the treatment of refractory benign esophageal strictures caused by caustic ingestion.
  Interventions: Device: Metal Stent (WallFlex™ Esophageal RX)

INTERVENTIONS:
Device: Metal Stent (WallFlex™ Esophageal RX)
  Other Names: WallFlex™ Esophageal RX Fully Covered Stent

SUMMARY:
The purpose of this study is to establish clinical proof of concept of temporary indwell of the WallFlex™ Esophageal Fully Covered Metal Stent (FCMS) for the treatment of refractory benign esophageal strictures caused by caustic ingestion.

DETAILED DESCRIPTION:
The purpose of this study is to establish clinical proof of concept of temporary indwell of the WallFlex™ Esophageal Fully Covered Metal Stent (FCMS) for the treatment of refractory benign esophageal strictures caused by caustic ingestion. Also to collect data in support of a hypothesis required to prospectively document the safety and effectiveness of temporary indwell of the WallFlex™ Esophageal Fully Covered Metal Stent (FCMS) compared to repeated Bougie Dilation for the treatment of refractory benign esophageal strictures caused by caustic ingestion.

ELIGIBILITY:
Inclusion Criteria:

1. Availability of medical history pertaining to dysphagia score prior to and during the preceding SECSER.
2. Availability of patient history pertaining to weight prior to and at completion of SECSER.
3. Benign esophageal stricture caused by caustic ingestion 12 or more weeks prior to enrollment.
4. Single esophageal stricture or multiple esophageal stricture over a length < 6 cm.
5. Having completed the SECSER consisting of 3 dilations intended to reach 15 mm each, separated by 2 weeks, followed by 3 dilations intended to reach 15 mm each with steroid injections, separated by 2 weeks. The dilations may be performed using Bougie or balloon dilation at the discretion of the investigator.
6. Refractory stricture defined as recurrence of stricture with associated dysphagia within 6 months after completion of SECSER.
7. Dysphagia score of 2 (ability to swallow semi-solid foods), 3 (ability to swallow liquids only) or 4 (unable to swallow liquids) at baseline.
8. Unable to pass a standard endoscope (approximately 9.8 mm diameter).
9. Age 18 years or older.
10. Willing and able to comply with the study procedures and provide written informed consent to participate in the study.

Exclusion Criteria:

1. Stricture within 2 cm of the upper esophageal sphincter.
2. Concomitant Esophageal ulcerations.
3. Prior esophageal stent placements.
4. Concurrent gastric and/or duodenal obstruction.
5. Patients with prior full or partial gastrectomy.
6. Sensitivity to any components of the stent or delivery system.
7. Concurrent medical condition that would affect the investigator's ability to evaluate the patient's condition or could compromise patient safety.
8. Participation in a clinical trial evaluating an investigational device within 3 months prior to enrollment in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2015-03; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- India (2):
  - Postgraduate Institute of Medical Education and Research, Chandigarh
  - Asian Institute of Gastroenterology, Hyderabad

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twenty (20) patients with refractory benign esophageal strictures caused by caustic ingestion were planned to be enrolled at 2-4 centers in India.
  * Group 1: Patients 1-10, stent indwell for 8 weeks +/- 7 days.
  * Group 2: Patients 11-20, stent indwell for 12 weeks +/- 7 days.
Groups:
- Metal Stent 8 Week Indwell: Patients 1 to 10 were to receive the WallFlex Esophageal Fully Covered Self-Expanding Metal Stent with stent indwell for 8 weeks +/- 7 days
- Metal Stent 12 Week Indwell: Patients 11 to 20 were to receive the WallFlex Esophageal Fully Covered Self-Expanding Metal Stent with stent indwell for 12 weeks +/- 7 days
Period: Overall Study
Arm/Group | Metal Stent 8 Week Indwell | Metal Stent 12 Week Indwell
Started (Patients 1-10, stent indwell for 8 weeks +/- 7 days.) | 1 | 0
Completed | 1 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | Metal Stent 8 Week Indwell
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: Years] | 54 [54 to 54]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Region of Enrollment [Number; unit: participants]
  India | 1

OUTCOME MEASURES:

1. Primary Outcome: Clinical Success
Description: Clinical success consisting of stent tolerability and adequate ability to sustain nutrition to 6 months after stent removal. Stent tolerability defined as absence of pain-related stent removal. Adequate ability to sustain nutrition defined as absence of dysphagia-related reintervention.
Time Frame: From stent placement on day 0 to 6 months after stent removal
Measure: Count of Participants; unit: Participants
Groups:
- Metal Stent 8 Week Indwell: The WallFlex™ Esophageal Fully Covered Metal Stent (FCMS) is being evaluated for the treatment of refractory benign esophageal strictures caused by caustic ingestion.
  Metal Stent (WallFlex™ Esophageal RX)
Arm/Group | Metal Stent 8 Week Indwell
Number analyzed (Participants) | 1
Participants | 1

2. Secondary Outcome: Stent Placement Success
Description: Number of participants with successful stent placement. Successful stent placement defined as the ability to deploy the stent in satisfactory position across the stricture
Time Frame: Stent placement on Day 0
Measure: Count of Participants; unit: Participants
Groups:
- Metal Stent 8 Week Indwell: The WallFlex™ Esophageal Fully Covered Metal Stent (FCMS)is being evaluated for the treatment of refractory benign esophageal strictures caused by caustic ingestion.
  Metal Stent (WallFlex™ Esophageal RX)
Arm/Group | Metal Stent 8 Week Indwell
Number analyzed (Participants) | 1
Participants | 1

3. Secondary Outcome: Stent Removal Success
Description: Number of participants with successful stent removal. Successful stent removal defined as the ability to remove the stent endoscopically without serious stent removal related complications.
Time Frame: Stent removal at Week 8 (±7 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Metal Stent 8 Week Indwell
Number analyzed (Participants) | 1
Participants | 1

4. Secondary Outcome: Change in Patient's Report on Pain Compared to Baseline
Description: Change in Patient's report on pain compared to Baseline at Day 2, Week 1, Week 2, Week 4, Week 6, and Thereafter every 2 weeks until stent removal at Week 8. Pain is reported on the VAS Pain Score scale from 0 (0 being No Pain) to 10 (10 being Worst Pain Ever). Higher score means a worse outcome.
  If reporting a score on a scale, please include the unabbreviated scale title, the minimum and maximum values, and whether higher scores mean a better or worse outcome.
Time Frame: From baseline to stent removal at Week 8 (±7 days)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Metal Stent 8 Week Indwell
Number analyzed (Participants) | 1
score on a scale
  Day 2 vs Baseline | 0
  Week 1 vs Baseline | 1
  Week 2 vs Baseline | 0
  Week 4 vs Baseline | 1
  Week 6 vs Baseline | 1
  Week 8 vs Baseline | 0

5. Secondary Outcome: Change of Pain Medication Intake From Baseline
Description: Change of pain medication intake from baseline at Day2, Week1, Week2, and thereafter every 2 weeks until stent removal
Time Frame: From baseline to stent removal at Week 8 (±7 days)
Population: Pain medication intake data not collected
Arm/Group | Metal Stent 8 Week Indwell
Number analyzed (Participants) | 0

6. Secondary Outcome: Change in Dysphagia Score Compared to Baseline
Description: Change in dysphagia score compared to Baseline at Day 2, Week 1, Week 2, Week 4, Week 6, Week 8, and thereafter every 2 weeks until end of study at Week 32. Change value was calculated as dysphagia score measured during stent treatment minus dysphagia score at Baseline.
  Dysphagia is reported using Dysphagia Scoring System (see scoring system below) with higher score meaning a worse outcome.
  0 = ability to eat a normal diet
  1. = ability to eat some solids
  2. = ability to eat some semisolids only
  3. = ability to swallow liquids only
  4. = complete dysphagia
Time Frame: From stent placement on day 0 to end of study at Week 32.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Metal Stent 8 Week Indwell
Number analyzed (Participants) | 1
Score on a scale
  Day2 vs Baseline | 0
  Week 1 vs Baseline | 0
  Week 2 vs Baseline | 0
  Week 4 vs Baseline | 0
  Week 6 vs Baseline | 0
  Week 8 vs Baseline | 0
  Week 10 vs Baseline | 0
  Week 12 vs Baseline | 0
  Week 14 vs Baseline | -1
  Week 16 vs Baseline | -1
  Week 18 vs Baseline | -1
  Week 20 vs Baseline | -1
  Week 22 vs Baseline | -1
  Week 24 vs Baseline | -1
  Week 26 vs Baseline | -1
  Week 28 vs Baseline | -1
  Week 30 vs Baseline | -1
  Week 32 vs Baseline | -1

7. Secondary Outcome: Dysphagia Score During Stent Treatment Compared to Score During Proceeding Standardized Esophageal Caustic Stricture Endoscopic Treatment Regimen (SECSER)
Description: Change in Dysphagia score during stent treatment compared to dysphagia score during proceeding standardized esophageal caustic stricture endoscopic treatment regimen (SECSER). Change value was calculated as dysphagia score during stent treatment (Day 2, Week 1, Week 2, and thereafter every 2 weeks until end of study at Week 32 minus dysphagia score at SECSER.
  Dysphagia is reported using Dysphagia Scoring System (see scoring system below) with higher score meaning a worse outcome.
  0. = ability to eat a normal diet
  1. = ability to eat some solids
  2. = ability to eat some semisolids only
  3. = ability to swallow liquids only
  4. = complete dysphagia
Time Frame: Dysphagia score at SECSER was measured prior to baseline. Dysphagia score during stent treatment was measured from stent placement on day 0 to end of study at Week 32
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Metal Stent 8 Week Indwell
Number analyzed (Participants) | 1
Score on a scale
  Day2 vs SECSR | -1
  Week 1 vs SECSR | -1
  Week 2 vs SECSR | -1
  Week 4 vs SECSR | -1
  Week 6 vs SECSR | -1
  Week 8 vs SECSR | -1
  Week 10 vs SECSR | -1
  Week 12 vs SECSR | -1
  Week 14 vs SECSR | -2
  Week 16 vs SECSR | -2
  Week 18 vs SECSR | -2
  Week 20 vs SECSR | -2
  Week 22 vs SECSR | -2
  Week 24 vs SECSR | -2
  Week 26 vs SECSR | -2
  Week 28 vs SECSR | -2
  Week 30 vs SECSR | -2
  Week 32 vs SECSR | -2

8. Secondary Outcome: Change in Quality of Life (QOL) Compared to Baseline
Description: Change in overall Quality of Life (QOL) health score compared to Baseline at Day 2, Week 1, Week 2, Week 4, Week 6, Week 8, and thereafter every 2 weeks until end of study at Week 32. QOL Overall Health Score is measured on a scale of 0 to 100, with 0 meaning the worst health you can imagine and 100 meaning the best health you can imagine. Higher score means a better outcome.
Time Frame: From stent placement on Day 0 to end of study at Week 32
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Metal Stent 8 Week Indwell
Number analyzed (Participants) | 1
Score on a scale
  Day 2 vs Baseline | 5
  Week 1 vs Baseline | 10
  Week 2 vs Baseline | 20
  Week 4 vs Baseline | 10
  Week 6 vs Baseline | 10
  Week 8 vs Baseline | 10
  Week 10 vs Baseline | 10
  Week 12 vs Baseline | 10
  Week 14 vs Baseline | 10
  Week 16 vs Baseline | 10
  Week 18 vs Baseline | 10
  Week 20 vs Baseline | 10
  Week 22 vs Baseline | 10
  Week 24 vs Baseline | 10
  Week 26 vs Baseline | 10
  Week 28 vs Baseline | 10
  Week 30 vs Baseline | 10
  Week 32 vs Baseline | 10

9. Secondary Outcome: Occurrence of Adverse Events
Description: Occurrence of Adverse Events Related to the Stent and/or the Stent Placement or Stent Removal Procedure and of All Serious Adverse Events Throughout the Duration of the Study
Time Frame: From stent placement on Day 0 to end of study at Week 32.
Measure: Number; unit: Adverse events
Arm/Group | Metal Stent 8 Week Indwell
Number analyzed (Participants) | 1
Adverse events | 0

10. Secondary Outcome: Time to Recurrence of Stricture
Description: Time to Recurrence of Stricture, Defined as Inability of a Normal Diameter Gastroscope (9.8 mm) to Pass the Stricture
Time Frame: From stent placement on Day 0 to end of study at Week 32.
Population: No recurrence of stricture
Arm/Group | Metal Stent 8 Week Indwell
Number analyzed (Participants) | 0

11. Secondary Outcome: Number of Stent Migration With or Without Related Adverse Events
Description: Number of stent migration with or without Related adverse events (AE). Stent migration is defined as any proximal or distal migration of stent.
Time Frame: From stent placement on Day 0 to end of study at Week 32.
Measure: Number; unit: Stent migrations
Arm/Group | Metal Stent 8 Week Indwell
Number analyzed (Participants) | 1
Stent migrations | 0

12. Secondary Outcome: Change in Patient Weight Compared to Baseline
Description: Change in Patient Weight Compared to Baseline: Day 2, Week 1, Week 2, Week 4, Week 6, Week 8, and Thereafter Every 2 Weeks Until End of Study at Week 32. Positive value means increase in weight and negative value means decrease in weight.
Time Frame: From stent placement on Day 0 to end of study at Week 32.
Measure: Number; unit: Kg
Arm/Group | Metal Stent 8 Week Indwell
Number analyzed (Participants) | 1
Kg
  Day 2 vs Baseline | 0
  Week 1 vs Baseline | -1
  Week 2 vs Baseline | -1
  Week 4 vs Baseline | -1
  Week 6 vs Baseline | -1
  Week 8 vs Baseline | 0
  Week 10 vs Baseline | -1
  Week 12 vs Baseline | -1
  Week 14 vs Baseline | -1
  Week 16 vs Baseline | -1
  Week 18 vs Baseline | -1
  Week 20 vs Baseline | 0
  Week 22 vs Baseline | 0
  Week 24 vs Baseline | -1
  Week 26 vs Baseline | -1
  Week 28 vs Baseline | -1
  Week 30 vs Baseline | -1
  Week 32 vs Baseline | -1

13. Secondary Outcome: Change in Patient Weight During Stent Treatment Compared to Weight Gain During Preceding SECSER
Description: Change in patient weight during stent treatment (day 2, week 1, week 2, week 4, week 6, week 8, and thereafter every 2 weeks until end of study at week 32) compared to preceding standardized esophageal caustic stricture endoscopic treatment regimen (SECSER). Positive value means increase in weight and negative value means decrease in weight.
Time Frame: From stent placement on Day 0 to end of study at Week 32.
Measure: Number; unit: kg
Arm/Group | Metal Stent 8 Week Indwell
Number analyzed (Participants) | 1
kg
  Day2 vs SECSR | 1
  Week 1 vs SECSR | 0
  Week 2 vs SECSR | 0
  Week 4 vs SECSR | 0
  Week 6 vs SECSR | 0
  Week 8 vs SECSR | 1
  Week 10 vs SECSR | 0
  Week 12 vs SECSR | 0
  Week 14 vs SECSR | 0
  Week 16 vs SECSR | 0
  Week 18 vs SECSR | 0
  Week 20 vs SECSR | 1
  Week 22 vs SECSR | 1
  Week 24 vs SECSR | 0
  Week 26 vs SECSR | 0
  Week 28 vs SECSR | 0
  Week 30 vs SECSR | 0
  Week 32 vs SECSR | 0

ADVERSE EVENTS:
Time Frame: Through completion of study at 32 weeks
Arm/Group | Metal Stent 8 Week Indwell
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days